CLINICAL TRIAL: NCT04574167
Title: Effects of tDCS Paired With Cognitive Training on Brain Networks Associated With Alcohol Use Disorder in Veterans
Acronym: tDCS/AUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBB-011-19S; VAM-19-00460 (Other: Minneapolis Veterans Affairs Medical Center); 1594744 (Other: IRBNet)
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: This study will be a double-blind, randomized, placebo (sham) controlled study of Veterans with AUD who will receive cognitive training and be randomized to either active or sham tDCS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Following enrollment in the study, participants will be randomized to either active or sham tDCS. Random permuted blocks will be used to ensure equal treatment numbers at certain equally-spaced points in the sequence of participant assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- tDCS with Cognitive Training (Experimental): Participants will receive 10 sessions of cognitive training concurrent with transcranial direct current stimulation (anode over left frontal cortex, cathode over right frontal cortex; 2 mAmps for 20 minutes)
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS with Cognitive Training (Sham Comparator): Participants will receive 10 sessions of cognitive training concurrent with sham tDCS. For sham tDCS, electrodes are placed at the same locations as for active tDCS, but current is ramped up for the initial 30 secs, then immediately ramped back down. This method mimics the initial physical sensation of stimulation, but there is no active current for the remainder of the session.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation (tDCS) — Cognitive training concurrent with 2 mAmps of anodal stimulation applied to the left frontal cortex for 20 minutes.
  Arms: tDCS with Cognitive Training
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Cognitive training concurrent with sham tDCS (30 secs ramp up/ramp down of current at beginning and end of session).
  Arms: Sham tDCS with Cognitive Training

SUMMARY:
Alcohol misuse is an epidemic among Veterans in the United States. Nearly 1/3 of Veterans have a lifetime history of Alcohol Use Disorder (AUD). In 2014, there were 15,306 unique patients treated in inpatient VA treatment programs alone, which represents a 10.7% increase from just two years prior. Unfortunately, about 2/3 of those entering treatment will relapse within one year.

Cognitive impairments found in chronic alcohol use interfere with adaptive behavior needed for successful recovery. These cognitive impairments and their underlying neural substrates may provide promising new targets for interventions that can reduce relapse rates. Evidence suggests that cognitive training can improve cognition in individuals with AUD, strengthen neural networks mediating cognition, and improve treatment outcome. However, cognitive training is effort intensive, has small effect sizes, and may have limited durability. The primary objective of this study is to investigate if transcranial direct current stimulation (tDCS) can increase the effectiveness of cognitive training to enhance cognition in alcohol use disorder and improve treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe Alcohol Use Disorder, according to DSM-5 within 12 months of enrollment (Participants may have current comorbid drug use, but their primary substance use disorder (SUD) diagnosis needs to be alcohol use based on self-report.)
* Veterans receiving outpatient clinical care services through the MVAHCS
* Abstinent from alcohol use for at least one week prior to the baseline study visit (Visit 1) (i.e., not in acute withdrawal) (Abstinence will be determined primarily via self-report, supplemented by breathalyzer, and clinical judgment based on other available data [e.g., perusal of medical records which may include urine test results and reports from clinicians in the Addiction Recovery Services Intensive Outpatient Program]).
* Men and women 22-70 years of age
* In the medical opinion of the PI, has been on a stable dose of all prescription and non-prescription medications (except for PRN medication) for at least 30 days prior to the baseline visit (Visit 1)
* Capable and willing to provide voluntary informed consent, in the medical opinion of the PI

Exclusion Criteria:

* Presence of a medical, psychiatric, physical or non-physical disease, disorder, condition, injury, disability or pre-existent history such that study participation, in the opinion of the PI: (a) may pose a significant risk to the participant; (b) raises the possibility that the participant is unlikely to successfully complete all of the requirements of the study according to the study protocol; or (c) might adversely impact the integrity of the data or the validity of the study results.
* Cognitive impairment as indicated by a score lower than or equal to 20 on the Montreal Cognitive Assessment (MoCA) or determined by the PI's judgment
* Psychosis or mania within 30 days of enrollment, as determined by the PI, based on a psychiatric history and examination and/or a review of available medical records
* Participant answers YES to Question 3 and NO to Question 6 (Moderate Risk) or participant answers YES to Question 4, 5, or 6 (High Risk) on the Columbia-Suicide Severity Rating Scale (C-SSRS) Screen Version - Recent Contraindications for tDCS (e.g., metallic cranial plates/screws or implanted device, eczema or skin lesions on scalp, presence of pacemakers, cochlea implants, or metal implants (excluding standard orthodontic braces, fillings, etc.))
* Contraindications for MRI (e.g., unapproved metallic implants, pacemakers or any other implanted electrical device, shrapnel, metallic braces, non-removable body piercings, significant breathing or movement disorder, claustrophobia) as assessed by completing the UMN CMRR Subject Safety Screening Form
* A positive pregnancy test result in a woman of childbearing age/potential as agreed upon by the PI

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Differences in change in frontal-striatal functional connectivity | Change between baseline and post-intervention (3 week) follow-up
  Participants will complete MRI sessions on a 3T scanner located in the Center for Magnetic Resonance Research (CMRR) at the University of Minnesota. Participants will undergo resting-state MRI over a 12-minute scan in order to gather resting state functional connectivity (RSFC). Hierarchical linear models will examine differences in change in target engagement (frontal-striatal RSFC) between active and sham tDCS conditions.
Change in Trail Making Test (TMT) score | Change between baseline and post-intervention (3 week) follow-up; 1 and 2 months following intervention
  The TMT is a neuropsychological test of visual attention and task switching. The test consists of two parts in which the participant is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The test can provide information about visual search speed, scanning, speed of processing, mental flexibility and executive functioning.
Change in Stroop Color-Word Test (SCWT) score | Change between baseline and post-intervention (3 week) follow-up; 1 and 2 months following intervention
  The SCWT is a neuropsychological test of the ability to inhibit cognitive interference which occurs when the processing of a stimulus feature affects the simultaneous processing of another attribute of the same stimulus.
Change in binge drinking days per week as measured using the Timeline Followback questionnaire | Change between baseline and post-intervention (3 week) follow-up; 1 and 2 months following intervention
  The TLFB questionnaire measures substance use disorder severity. The questionnaire asks the participant about substance use in the past 30 days. The participant reports on a binary scale as to whether or not they have used a given substance. Binge drinking is defined as men consuming 5 or more drinks or women consuming 4 or more drinks in about 2 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin O Lim, MD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data may be shared upon request.

DOCUMENTS (1):
  • Informed Consent Form (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT04574167/ICF_000.pdf